CLINICAL TRIAL: NCT03309228
Title: Subjective Factors of Polymedication in the Elderly: a Qualitative Study of the Perceptions of Patients, Relatives and Referent Physicians.(DOSAGE)
Acronym: DOSAGE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Responsible Party: Sponsor
Other Study IDs: DOSAGE
Record Dates: First submitted 2017-10-10; First posted 2017-10-13 (Actual); Last update posted 2018-07-18 (Actual); Status verified 2017-10

CONDITIONS: Frail Elderly Syndrome
Keywords: elderly people; polymedication,; ethics; qualitative research

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Qualitative Research: Semi-structured interviews with patients, relatives and general practitioners.
  Interventions: Other: individual interviews

INTERVENTIONS:
Other: individual interviews — Semi-structured individual interviews with patients, relatives and general practitioners.

SUMMARY:
The DOSAGE Study is a qualitative transversal study aiming to describe and understand the subjective factors of polymedication in the elderly population (75 years old and more), defined as 10 simultaneous drugs. Semi-structured interviews will be conducted with patients, relatives and general practitioners in one French region. 20 situations will be included. After analysing the data of the individual interviews, focus groups will be conducted with health professionals.

ELIGIBILITY:
Inclusion Criteria:

* For patients:

  * Men and women aged 75 and over
  * Beneficiary of a prescription of medicinal products fulfilling the conditions of major polymedication: to include 10 different drugs whatever the way of use (per os, subcutaneous, intravenous, intra muscular, cutaneous, instillation)
  * Informed consent stating that the subject understood the purpose and methodology of the study and agrees to participate in the study.
* For the relatives:

  * Men and women 18 years of age or older
  * Informed consent
  * Regularly participating in helping the patient's daily life
* For Physicians :

  * Identified as the patient's physician or family physician.
  * Informed consent

Exclusion Criteria:

* Persons with proven and significant cognitive impairment preventing the completion of semi-strutured interviews
* Person who does not speak French easily
* Generally, any person unlikely to cooperate in the study
* Adults under guardianship
* Refusal of relatives and/or general practitioner to participate to the study

Min Age: 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: Men and women aged 75 and over, fulfilling the conditions of major polymedication: (10 different simultaneous drugs)
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2016-11-16 (Actual); Primary Completion 2019-11 (Estimated); Study Completion 2022-11 (Estimated)

PRIMARY OUTCOMES:
60 semi-structured interviews | 9 months
  Qualitative data analysis - Theorical saturation

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Besançon, Besançon, France

IPD SHARING:
Plan to Share IPD: No